CLINICAL TRIAL: NCT06320405
Title: A Phase Ib/II Study of Axatilimab in Combination With Retifanlimab and Paclitaxel for the Treatment of Patients With Advanced Solid Tumors
Brief Title: Axatilimab in Combination With Retifanlimab and Paclitaxel for the Treatment of Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Shivaani Kummar, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025940; NCI-2024-01397 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025940 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — axatilimab; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (axatilimab, retifanlimab, paclitaxel) (Experimental): Patients receive axatilimab IV over 30 minutes on day -8, prior to cycle 1. Beginning in cycle 1 day 1, patients receive axatilimab IV over 30 minutes on days 8 and 21 of each cycle, retifanlimab IV over 30-60 minutes on day 1 of each cycle, and paclitaxel IV over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy, CT scan, and blood sample collection throughout the study and may undergo MRI and/or PET scan throughout the study.
  Interventions: Biological: Axatilimab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Biological: Retifanlimab

INTERVENTIONS:
Biological: Axatilimab — Given IV
  Other Names: Anti-M-CSFR Monoclonal Antibody SNDX-6352; SNDX 6352; SNDX-6352; SNDX6352; UCB6352
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Retifanlimab — Given IV
  Other Names: INCMGA 0012; INCMGA-0012; INCMGA00012; INCMGA0012; MGA 012; MGA-012; MGA012; Retifanlimab-dlwr; Zynyz

SUMMARY:
This phase I/II trial tests the safety, side effects, and effectiveness of axatilimab in combination with retifanlimab and paclitaxel for the treatment of patients with a solid tumor that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Axatilimab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as retifanlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Giving axatilimab in combination with retifanlimab and paclitaxel may be safe, tolerable and/or effective in treating patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Phase Ib: Determine the safety and tolerability of the combination of axatilimab, retifanlimab, and paclitaxel in patients with advanced solid tumors.

II. Phase II: Determine the efficacy of the combination of axatilimab, retifanlimab, and paclitaxel in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of the combination of axatilimab, retifanlimab, and paclitaxel in patients with advanced solid tumors treated in phase II.

II. Explore treatment related changes in the tumor microenvironment (TME) following treatment with the combination of axatilimab, retifanlimab, and paclitaxel in advanced solid tumors.

III. Assess predictive biomarkers of response in peripheral blood.

OUTLINE:

Patients receive axatilimab intravenously (IV) over 30 minutes on day -8, prior to cycle 1. Beginning in cycle 1 day 1, patients receive axatilimab IV over 30 minutes on days 8 and 22 of each cycle, retifanlimab IV over 30-60 minutes on day 1 of each cycle, and paclitaxel IV over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy, computed tomography (CT) scan, and blood sample collection throughout the study and may undergo magnetic resonance imaging (MRI) and/or positron emission tomography (PET) scan throughout the study.

After completion of study treatment, patients are followed up at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the investigational nature of the study and provide informed consent. Written informed consent must be obtained prior to any study specific procedures or interventions
* Age ≥ 18 years at the time of consent. All participants, irrespective of their gender, gender identity, race, and ethnicity, will be included
* Certified, documented diagnosis of a metastatic solid tumor based on pathology review
* Presence of at least one lesion that is measurable per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and another lesion that is amenable to tumor biopsy
* Relapsed from, or refractory to, standard of care (SOC) systemic therapy known to prolong survival or if, in the opinion of the primary treating oncologist, a clinical trial is the best option for the next line of treatment based on response and/or tolerability to available therapies
* Investigational therapy is permitted after a wash-out period of 5 half-lives (if known), or 28 days, whichever is shorter, prior to study day -8. Prior use of an investigational agent for imaging, such as T cell imaging, is permitted
* Prior treatment with taxanes. A wash-out of period of ≥ 3 months prior to day -8 must be met for enrollment. Prior anti PD-1/PD-L1 therapy is allowed, but not required
* Eastern Cooperative Oncology Group (ECOG) status (performance status [PS]) of 0-1
* Life expectancy of greater than 12 weeks according to certified physician review
* Hemoglobin (Hb) ≥ 8.5 g/dL
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelets ≥ 100K/cc mL

  * Values must be obtained without transfusion within 2 weeks
* Serum creatinine (sCr) < 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 50 mL/min (calculated with the Cockcroft-Gault formula) for participants with creatinine (sCr) levels above institutional normal
* Total bilirubin < 1.5 x upper limit of normal (ULN)

  * With the exception of documented Gilbert's syndrome or similar conditions, at the discretion of the principal investigator (PI). Clinical chemistry testing may be adjusted, as clinically indicated
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Corrected QT interval Fridericia's formula (QTcF) of < 480 ms on a 12 lead electrocardiogram (EKG), except for participants with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid
* Willingness to modify concomitant drug regimens, at the recommendation and discretion of pharmacy services, including the use of known substrates or inhibitors of CYP2C8 and CYP3A4
* Physiologic maintenance doses of corticosteroids (≤ 10 mg/day of prednisone or equivalent) are permitted. Examples include: Asthma treatment; topical ocular, intra-articular, or intranasal steroids with minimal systemic absorption; and brief courses of corticosteroids for prophylaxis
* Patients with CD4+ T-cell (CD4+) counts ≥ 350 cells/uL are eligible regardless of HIV serology

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible
  * In the case of ongoing treatment with antiretroviral therapy (ART), medication adjustment may be necessary for the duration of treatment. A wash-out period may be necessary, at the recommendation of the institutional research pharmacy service (RPS)
* Evidence of chronic hepatitis B virus (HBV) infection (i.e., hepatitis B surface antigen [HBsAg]-positive, undetectable or low HBV deoxyribonucleic acid [DNA], and normal ALT) in the absence of HBV therapy, or serologic evidence of a resolved prior HBV infection (i.e., HBsAg-negative and hepatitis B virus core antibody [anti-HBc]-positive) is permitted
* History of hepatitis C virus (HCV) infection is permitted given prior curative treatment or undetectable HCV viral load by serology or polymerase chain reaction (PCR) testing

  * Patient who are HCV antibody (Ab) seropositive but HCV ribonucleic acid (RNA) negative due to prior treatment or natural resolution are eligible

Exclusion Criteria:

* Secondary malignancy with documented diagnosis by a treating physician < 3 years prior to study day -8. The following criteria also apply:

  * New or progressive brain metastases. Patients with brain metastases not requiring immediate central nervous system (CNS) specific treatment or stable for at least 4 weeks prior to study day -8 are eligible at the discretion of the investigator given that neurologic symptoms are resolved.
  * Patients with active leptomeningeal disease are not eligible
* Palliative radiation therapy administered within 1 week prior to study day -8, Note: Participants must have recovered from all radiation-related toxicities (to grade < 1 or baseline), must not require corticosteroids for this purpose, and must not have had radiation pneumonitis
* Immunization with a live vaccine within 28 days prior to study day -8
* History of organ transplantation, including hematopoietic stem cell transplantation (HSCT)
* Clinical evidence of interstitial lung disease or active non-infectious pneumonia
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (≤ 10 mg/day of prednisone or equivalent is permitted)
* Prior National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 immune-related adverse event (irAE) that required systemic immunosuppression (endocrinopathies managed by stable doses of supplements and/or corticosteroids ≤ 10 mg/day are permitted)
* Unresolved toxicities (resolution required to grade 1 or baseline) from prior anticancer therapies. The following exceptions apply:

  * Alopecia, lymphopenia, grade 2 neuropathy (if not resulting in functional deficit), and grade 1 (no supplementation required) or grade 2 endocrinopathies (stable on supplements)
* Prior allergy or severe hypersensitivity reaction to axatilimab, retifanlimab, paclitaxel, cremaphor-containing agents, and/or components of the drug formulations
* Active infection requiring systemic antibiotic therapy
* Persons of childbearing potential (PCBP) who are pregnant (i.e., positive pregnancy test within 7 days prior to study day -8) or breastfeeding are not eligible.

  * The effects of the investigational regimen on the developing human fetus are unknown. For this reason, persons of reproductive potential must agree to use a highly effective form of contraception, starting with the time of consent to 4 months after the last dose of retifanlimab or 90 days after the last dose of axatilimab, whichever is longer
  * Sperm-producing participants must not donate sperm throughout the study period and for 90 days post completion of study treatment
* Uncontrolled, intercurrent illness and psychiatric illness/social situations that would limit compliance with study requirements, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (phase Ib) | From the first dose of axatilimab (day -8) to the end of cycle 1 (cycle is 28 days starting from cycle 1 day 1 [first dose of retifanlimab and paclitaxel])
  Will be coded by system organ class, MedDRA preferred term, and severity grade using Common Terminology Criteria for Adverse Events (version 5.0).
Recommended phase 2 dose of the study drug combination (phase Ib) | From the first dose of axatilimab (day -8) to the end of cycle 1 (cycle is 28 days starting from cycle 1 day 1 [first dose of retifanlimab and paclitaxel])
Clinical benefit rate (phase Ib/II) | From screening assessment to the end of cycle 6 assessment (each cycle is 28 days starting from cycle 1 day 1 [first dose of retifanlimab and paclitaxel])
  Defined as percentage of participants with complete response or partial response confirmed by scans at least 4 weeks apart, or stable disease for > 4 months. Will be reported with exact 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of ≥ grade 3 toxicities possibly or definitely related to study drugs | From the first dose of axatilimab (day -8) to 90 days after the end of treatment visit (an average of 6 months)
  Will be categorized and tabulated for reporting. The analyses for reporting may include descriptive statistical analyses of the overall set of phase II adverse events.
Changes in immune cell composition and functionality | From screening until cycle 2 day 1 biopsy (each cycle is 28 days starting from cycle 1 day 1 [first dose of retifanlimab and paclitaxel])
  Will be characterized in peripheral blood using flow cytometry (FC) and candidate protein biomarkers will be identified in tumor tissue using multiplexed immunohistochemistry. Changes in immune cell composition and functionality at the biopsy during cycle 2 will be assessed by paired t-test.
Change in immune cell population | From screening to end of treatment visit (an average of 6 months)
  To assess predictive biomarkers of response in peripheral blood, changes in immune cell populations in peripheral blood, including reduced presence of CD14dimCD16+ monocytes and increased presence of CD8+ T effector memory subsets, at the end of the study between responders and non-responders will be assessed using repeated measures of analysis of covariance over time to accommodate a longitudinal nature of peripheral blood draws for flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States